CLINICAL TRIAL: NCT02814110
Title: Efficacy and the Safety of Granulocyte Colony-stimulating Factor Treatment in Children and Adolescents With Muscular Dystrophy: An Open Study
Brief Title: Efficacy Safety of Granulocyte Colony-stimulating Factor Treatment Children and Adolescents With Muscular Dystrophy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Bialystok (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMB 143-20899 P
Record Dates: First submitted 2016-06-23; First posted 2016-06-27 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Increase Muscle Strength in Patients With Muscular Dystrophy
Keywords: Granulocyte colony-stimulating factor; muscular dystrophy; muscle strength; children; adolescents
MeSH Terms: conditions — Muscular Dystrophies | interventions — Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Granulocyte colony-stimulating factor (Other): Granulocyte colony-stimulating factor Muscle strength Muscular dystrophy
  Interventions: Drug: Granulocyte colony-stimulating factor (Filgrastim)

INTERVENTIONS:
Drug: Granulocyte colony-stimulating factor (Filgrastim) — Drug administration
  Other Names: Filgrastim

SUMMARY:
Importance: Currently the gold standard treatment for ambulant patients is corticosteroids. Granulocyte colony-stimulating factor (G-CSF) has been reported to exert the proliferation of satellite cells, the regulation of myoblast proliferation, and the differentiation and promotion of muscle regeneration and repair.

Objectives To evaluate the safety and efficacy of G-CSF in children and adolescents with muscular dystrophies Duchenne muscular dystrophy, Becker muscular dystrophy , Fascioscapulohumeral dystrophy.

Design, Setting, and Participants: Patients aged 5-15 with diagnosed muscular dystrophies will be included in an open study. Patients wheelchair-bound and and mobile and self-independent can participate in the study. Patients also treated with steroids can participate in this study. Clinical examination and physiotherapeutic and laboratory tests will be perform. G-CSF (5mcg/kg/body/d) is given subcutaneously for five consecutive days during the 1st, 2nd, 3rd. 6th and 12th months. Manual muscle testing (Lovett test) of the upper and lower extremities, isometric force with the hand dynamometer, and the 6MWT (six minute walk test) are measured before and after therapy.

DETAILED DESCRIPTION:
Importance: Currently the gold standard treatment for ambulant patients is corticosteroids. Granulocyte colony-stimulating factor (G-CSF) has been reported to exert the proliferation of satellite cells, the regulation of myoblast proliferation, and the differentiation and promotion of muscle regeneration and repair.

Objectives To evaluate the safety and efficacy of G-CSF in children and adolescents with muscular dystrophies Duchenne muscular dystrophy, Becker muscular dystrophy , Fascioscapulohumeral dystrophy.

Design, Setting, and Participants: Patients aged 5-15 with diagnosed muscular dystrophies will be included in an open study. Patients wheelchair-bound and and mobile and self-independent can participate in the study. Patients also treated with steroids can participate in this study. Clinical examination and physiotherapeutic and laboratory tests will be perform. G-CSF (5mcg/kg/body/d) is given subcutaneously for five consecutive days during the 1st, 2nd, 3rd. 6th and 12th months. Blood is sampled before G-CSF administration and on the 5th day of each treatment cycle.

During each cycle of G-CSF administration physical therapy is also applied. Abdominal ultrasonography with a spleen assessment is performed before and after 7 days of G-CSF administration. Spirometry and electrocardiographic record are also performed. Side effects of G-CSF treatment will be assessed.

Manual muscle testing (Lovett test) of the upper and lower extremities, isometric force with the hand dynamometer, and the 6MWT (six minute walk test) are measured before and after therapy. MRI of the gastrocnemius muscles will performed at the beginning and at the end of therapy.

ELIGIBILITY:
Inclusion Criteria:

* Muscular dystrophy - Duchenne muscular dystrophy, Becker muscular dystrophy, Fascioscapulohumeral dystrophy
* age 5-15

Exclusion Criteria:

* non- muscular dystrophy
* age below 5 years
* age over 15 years

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 27 (Estimated)
Dates: Start 2013-03-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety based on number of participants with adverse events. | Seven years
  Adverse events will be monitored and scored for severity and related to the Granulocyte Colony-Stimulating Factor administration.

SECONDARY OUTCOMES:
Muscle strength in patients with muscular dystrophy | Seven years
  The assessment of muscle strength of the upper and lower limbs by Lovett test. The evaluation isometric force of upper limbs with the hand dynamometer.
  Distance measurement in a 6-minute walk test (6MWT) by feet or wheelchair,6MWT before and after therapy.
Laboratory investigations in patients with muscular dystrophy | Seven years
  Blood count: Red blood cells 10^6/µL; Hemoglobin g/dl, Leucocytes 10^3/µL, Platelets 10^3/µL; biochemistry CRP - C Reactive Protein - mg/L; creatinine - mg/dL; glucose mg/dL, electrolytes, AST- U/L; ALT - U/L; cholesterol mg/dL; fibrinogen - mg/dL, partial thromboplastin time - sec; prothrombin time - sec, creatine kinase - U/L
Abdominal ultrasonography in patients with muscular dystrophy | Seven years
  Abdominal ultrasonography with a spleen measurement will be done before and after G-CSF administration
Electrocardiographic records in patients with muscular dystrophy | Seven years
  Electrocardiographic records wiil ibe done in patients with muscular Dystrophy before and after G-CSF administration.

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Kulak, MD,PhD,Prof, Principal Investigator — Medical University of Bialystok, Bialystok, Poland
Locations (1):
- Department of Pediatric Rehabilitation, Bialystok, Podlaskie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sienkiewicz D, Kulak W, Paszko-Patej G, Okurowska-Zawada B, Sienkiewicz J, Kulak P. Biochemical Changes in Blood of Patients with Duchenne Muscular Dystrophy Treated with Granulocyte-Colony Stimulating Factor. Biomed Res Int. 2019 Mar 13;2019:4789101. doi: 10.1155/2019/4789101. eCollection 2019. PMID 31001554
- [Result] Sienkiewicz D, Kulak W, Okurowska-Zawada B, Paszko-Patej G, Wojtkowski J, Sochon K, Kalinowska A, Okulczyk K, Sienkiewicz J, McEachern E. Efficacy and the Safety of Granulocyte Colony-Stimulating Factor Treatment in Patients with Muscular Dystrophy: A Non-Randomized Clinical Trial. Front Neurol. 2017 Oct 26;8:566. doi: 10.3389/fneur.2017.00566. eCollection 2017. PMID 29123500
- [Result] Eljaszewicz A, Sienkiewicz D, Grubczak K, Okurowska-Zawada B, Paszko-Patej G, Miklasz P, Singh P, Radzikowska U, Kulak W, Moniuszko M. Effect of Periodic Granulocyte Colony-Stimulating Factor Administration on Endothelial Progenitor Cells and Different Monocyte Subsets in Pediatric Patients with Muscular Dystrophies. Stem Cells Int. 2016;2016:2650849. doi: 10.1155/2016/2650849. Epub 2015 Dec 6. PMID 26770204